CLINICAL TRIAL: NCT05511571
Title: The Effect of Progressive Relaxation Exercises and Transcutaneous Electrical Nerve Stimulation Administered to Women Delivering Via Cesarean Section on Acute Pain, Breastfeeding Behaviors, and Comfort Levels: A Randomized Controlled Study
Brief Title: Effect of Progressive Relaxation Exercises and TENS on Women Delivering Via Cesarean
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Derya Öztürk Özen (Other)
Collaborators: Hacettepe University (Other); Saglik Bilimleri Universitesi (Other)
Responsible Party: Sponsor-Investigator, Derya Öztürk Özen, Principal Investigator, Bozok University
Organization: Bozok University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: KA-17142
Record Dates: First submitted 2022-08-17; First posted 2022-08-23 (Actual); Last update posted 2022-08-23 (Actual); Status verified 2022-08

CONDITIONS: Cesarean Section; Acute Pain
Keywords: cesarean section; pain; breastfeeding; comfort; muscle relaxation; transcutaneous electrical neural stimulation
MeSH Terms: conditions — Acute Pain; Pain; Breast Feeding | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- TENS group (Experimental): Transcutaneous electrical neural stimulation (TENS)
  Interventions: Device: Transcutaneous electrical neural stimulation (TENS)
- PRE group (Experimental): Progressive relaxation exercises (PRE)
  Interventions: Other: Progressive relaxation exercises (PRE)
- TENS+PRE group (Experimental): Transcutaneous electrical neural stimulation (TENS) and Progressive relaxation exercises (PRE)
  Interventions: Other: Transcutaneous electrical neural stimulation (TENS) and Progressive relaxation exercises (PRE)
- Control group (No Intervention)

INTERVENTIONS:
Device: Transcutaneous electrical neural stimulation (TENS) — The TENS group: TENS application was implemented by the researchers in the patient room. The conventional TENS application took 30 minutes per session. The application continued until frequency reached 100 Hz, the pulse width reached 100 μs, and the current impedance reached a point where the women felt needling or tingling according to their tolerance. Before the application, the women were asked to lie in a supine position, and the area/skin where TENS would be applied was cleaned and dried. Two electrodes of TENS were placed 2 cm above the cesarean incision, and the other two electrodes 2 cm below the incision. The women were allowed to rest during the application, and they were accompanied by the researcher. A total of five TENS sessions, including two at four-hour intervals on the first day and three at eight-hour intervals on the second day, were held.
  Arms: TENS group
Other: Progressive relaxation exercises (PRE) — The PRE group: The PRE application was implemented in the patient room. A quiet and calm environment was prepared in the room for the intervention. The PRE application was implemented by the women under the researchers' instructions. Each session lasted 30 minutes. A total of five sessions, including two at four-hour intervals on the first day and three at eight-hour intervals on the second day, were held. The PRE application includes exercises based on stretching and then the relaxation of different muscle groups, accompanied by deep breathing. The exercises were carried out in the following way: First doing a deep breathing exercise and then stretching all the muscles from feet to face accompanied by breathing in, keeping the breath, and finally relaxing the muscles by breathing out at the same time.
  Arms: PRE group
Other: Transcutaneous electrical neural stimulation (TENS) and Progressive relaxation exercises (PRE) — The TENS+PRE group: The PRE and TENS applications were carried out together in this group. The administration of the interventions was the same as in groups where only TENS and only PRE applications were carried out. In this group, first, a 30-minute PRE application was implemented, which was followed by a 30-minute-TENS application.
  Arms: TENS+PRE group

SUMMARY:
This study aimed to determine the effect of progressive relaxation exercises and transcutaneous electrical nerve stimulation administered to women delivering via cesarean section on acute pain, breastfeeding behavior, and comfort levels. Single-Blind, Randomized Controlled Study. This study was carried out in the obstetrics and gynecology clinic of a university hospital affiliated with the Ministry of Health in Turkey between August 20, 2018 and April 15, 2019. A total of 120 participants were randomly assigned to one of four groups, which included a transcutaneous electrical neural stimulation (TENS) group, a progressive relaxation exercises (PRE) group, a combined intervention (TENS+PRE) group, and a control group. Data were collected with a data collection form, the visual analogue scale (VAS), the LATCH breastfeeding diagnostic tool (LATCH), and the postpartum comfort scale (PCS). In the analysis of the data, numbers, percentages, and chi-square tests were used. Also, median values, Wilcoxon Signed-rank test, and Kruskal-Wallis H test were employed for continuous variables.

ELIGIBILITY:
Inclusion Criteria:

* women who were aged between 18 and 45,
* who were in the postoperative 8th hour,
* who had a transverse cesarean section,
* who, as well as their babies, did not develop any complications during pregnancy, delivery, and the postpartum period.

Exclusion Criteria:

* women who did not have an open wound on their body and/or allergic disease on their skin,
* who had cardiac arrhythmia or a pacemaker,
* who had a risk of epilepsy,
* who had epilepsy, eclampsia, kidney or liver disease,
* who had previously applied TENS and PRE methods,
* who were morbidly obese (with a BMI value of over 40),
* who used chronic opioids, antidepressants, and psychoactive drugs.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2018-08-20 (Actual); Primary Completion 2019-04-15 (Actual); Study Completion 2019-04-15 (Actual)

PRIMARY OUTCOMES:
Change in acute pain | VAS was applied in the first eighth hour during the postoperative 48 hours, before and after each application in the intervention groups, and in the control group at the times corresponding to the applications in the intervention groups.
  The Visual Analog Scale (VAS) was used in the evaluation of acute pain.

SECONDARY OUTCOMES:
Change in breastfeeding behavior | LATCH was applied in the first eighth hour (before the first application) during the postoperative 48 hours. It was applied again on the first and second days when all interventions were completed.
  The LATCH Breastfeeding Diagnostic Tool (LATCH) was used in the evaluation of breastfeeding behavior.
Change in comfort level | Postpartum Comfort Scale was applied in the first eighth hour (before the first application) during the postoperative 48 hours. It was applied again on the first and second days when all interventions were completed.
  The Postpartum Comfort Scale was used in the evaluation of comfort level.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Health Sciences, Ankara, Turkey (Türkiye)